CLINICAL TRIAL: NCT03657355
Title: Randomized, Double-blind, Double-dummy, Placebo- and Active-controlled, 6-way Cross-over Study to Evaluate the Abuse Potential of Single, Oral Doses of ACT-541468 in Healthy Recreational Drug Users
Brief Title: Study to Evaluate the Abuse Potential of ACT-541468 in Healthy Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078-107
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Healthy Recreational Drug Users
MeSH Terms: interventions — daridorexant; suvorexant; Zolpidem

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, double-dummy, placebo- and active-controlled, 6-way cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For blinding purposes, suvorexant and zolpidem will be over-encapsulated, whereas a matching-placebo will be used for ACT-541468.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 50 mg ACT-541468 (Experimental): ACT-541468 will be administered as tablets for oral use.
  Interventions: Drug: ACT-541468
- 100 mg ACT-541468 (Experimental): ACT-541468 will be administered as tablets for oral use.
  Interventions: Drug: ACT-541468
- 150 mg ACT-541468 (Experimental): ACT-541468 will be administered as tablets for oral use.
  Interventions: Drug: ACT-541468
- 150 mg suvorexant (Active Comparator): Suvorexant will be administered as tablets for oral use.
  Interventions: Drug: Suvorexant
- 30 mg zolpidem (Active Comparator): Zolpidem will be administered as tablets for oral use.
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator): Placebo will be administered as tablets for oral use.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-541468 — ACT-541468 will be administered as 50 mg tablets for oral use.
  Arms: 100 mg ACT-541468; 150 mg ACT-541468; 50 mg ACT-541468
Drug: Suvorexant — Suvorexant will be administered as 15 mg over-encapsulated tablets for oral use.
  Arms: 150 mg suvorexant
Drug: Zolpidem — Zolpidem will be administered as 10 mg over-encapsulated tablets for oral use.
  Arms: 30 mg zolpidem
Drug: Placebo — Matching-placebo will be used.
  Arms: Placebo

SUMMARY:
This placebo- and active controlled study will investigate the abuse potential of ACT-541468 in healthy recreational drug users

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Male or female healthy subjects, 18-55 years of age (inclusive) at Screening
* Body mass index of 18.0-33.0 kg/m2 (inclusive) at Screening and a minimum weight of 50.0 kg at Screening
* Current sedative users who have used sedatives (e.g., benzodiazepines, zolpidem, eszopiclone, gamma-hydroxybutyrate, barbiturates) for recreational (non-therapeutic) purposes (i.e., for psychoactive effects) at least ten times in their life and at least once in the 12 weeks before Screening
* Women of childbearing potential must consistently and correctly use a reliable method of contraception with a failure rate of < 1% per year, be sexually inactive, or have a vasectomized partner
* Women of non-childbearing potential
* Male subjects are required to use a medically acceptable method of contraception throughout the entire study period and for at least 90 days after last study drug administration

Exclusion Criteria:

* History of major medical or surgical disorders which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment(s)
* Positive HIV or hepatitis B/C test at Screening
* Female subjects who are currently pregnant or lactating or who are planning to become pregnant within 1 month of the last study treatment administration
* Modified Swiss Narcolepsy Scale total score < 0 at Screening or history of narcolepsy or cataplexy
* Substance or alcohol dependence within 2 years prior to Screening or prior participation in a substance or alcohol dependence rehabilitation program
* Subjects who have a positive urine drug screen at admittance to the qualification or core phase
* Any sleep-disorder including self-reported insomnia disorder, breathing-related sleep disorders, restless legs syndrome (RLS), nightmare disorder, non-rapid eye movement (REM), sleep arousal disorders, REM sleep behavior disorder, circadian rhythm sleep-wake disorders, or narcolepsy
* Any of the following SLEEP-50 Questionnaire scores at Screening:

  * ≥ 15 on Apnea subscale;
  * ≥ 7 on Narcolepsy subscale;
  * ≥ 7 on RLS or Periodic limb movement disorder subscale;
  * ≥ 8 on Circadian Rhythm subscale;
  * ≥ 7 on Sleepwalking subscale;
  * ≥ 3 on Item 32 and ≥ 9 on Items 33 to 35 (i.e., on nightmare subscale);
  * ≥ 15 on Impact subscale.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Maximum effect (Emax) of the Drug Liking VAS ('at this moment') over 24 h post-dose during each treatment period | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale

SECONDARY OUTCOMES:
Drug Liking VAS (bipolar) | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale
Overall Drug Liking VAS (bipolar) | Duration: for up to 12 hours post-dose
  VAS = visual analogue scale
Take Drug Again VAS (bipolar) | Duration: for up to 12 hours post-dose
Good Effects VAS (unipolar) | Duration: for up to 24 hours post-dose
Drug Similarity VAS | Duration: for up to 1 hour post-dose
  VAS = visual analogue scale
Bad Effects VAS (unipolar) | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale
Alertness/Drowsiness VAS (bipolar) | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale
Any Effects VAS (unipolar) | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale
Feeling High VAS (unipolar) | Duration: for up to 24 hours post-dose
  VAS = visual analogue scale
Bowdle VAS Internal and External Perceptions | Duration: for up to 24 hours post-dose
Observer's Assessment of Alertness/Sedation composite and sum scores | Duration: for up to 24 hours post-dose
Reaction time task score | Duration: for up to 8 hours post-dose
Rapid visual information processing score | Duration: for up to 8 hours post-dose
Paired Associates Learning score | Duration: for up to 8 hours post-dose

OTHER OUTCOMES:
AUC(0-t) of ACT-541468 | Duration: for up to 24 hours post-dose
AUC(0-∞) of ACT-541468 | Duration: for up to 24 hours post-dose
Cmax of ACT-541468 | Duration: for up to 24 hours post-dose
tmax of ACT-541468 | Duration: for up to 24 hours post-dose
t½ of ACT-541468 | Duration: for up to 24 hours post-dose
Treatment-emergent adverse events (AEs) | All AEs from (first) admittance on Day -1 up to EOS, i.e. for up to 9 weeks
Treatment-emergent serious AEs (SAEs) | SAE reporting: from signature of informed consent up to EOS, i.e. for up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (2):
- Altasciences Clinical Kansas, Inc. (former Vince and Associates Clinical Research, Inc.), Overland Park, Kansas, United States
- Altasciences Company Inc., Montreal, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ufer M, Kelsh D, Schoedel KA, Dingemanse J. Abuse potential assessment of the new dual orexin receptor antagonist daridorexant in recreational sedative drug users as compared to suvorexant and zolpidem. Sleep. 2022 Mar 14;45(3):zsab224. doi: 10.1093/sleep/zsab224. PMID 34480579